CLINICAL TRIAL: NCT00146835
Title: Phase IV, Prospective Study of the Safety of GSK Bios' Pediarix Administered to a Cohort of Infants in a US Health Maintenance Organization (HMO). (Post-Marketing PEDIARIX Safety Study)
Brief Title: Post-marketing Safety Study of GSK Biological's Pediarix™ Vaccine
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Kaiser Permanente (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: 217744/088
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Hepatitis B; Poliomyelitis; Diphtheria; Tetanus; Acellular Pertussis
MeSH Terms: conditions — Hepatitis B; Poliomyelitis; Diphtheria; Tetanus | interventions — PEDIARIX; Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Cohort A: The primary study cohort includes all infants from SCKP who have begun their primary course of vaccine with PEDIARIX co-administered with Prevnar and for whom at least one dose of PEDIARIX was administered prior to the infant's 9-month birthday and safety follow-up information is available.
  Interventions: Biological: Pediarix; Biological: Prevnar®: (Wyeth)
- Cohort B: This Historical cohort includes age-, gender- and area-matched infants who received at least one dose of DTaP vaccine co-administered with 7Pn between 1 January 2002 and 29 April 2003.
  Interventions: Biological: Licensed DTPa containing vaccine; Biological: Prevnar®: (Wyeth)
- Cohort C: This "delayed Pediarix use clinics" cohort includes all infants who, during the enrollment period for Cohort A, begin their primary course of vaccination with a DTaP vaccine co-administered with 7Pn. It is age-, gender-, and area-matched in a similar manner to Cohort B.
  Interventions: Biological: Licensed DTPa containing vaccine; Biological: Prevnar®: (Wyeth)

INTERVENTIONS:
Biological: Pediarix — 1 or more injections
  Groups: Cohort A
Biological: Licensed DTPa containing vaccine — 1 or more injections
  Groups: Cohort B; Cohort C
Biological: Prevnar®: (Wyeth) — Concomitant vaccination

SUMMARY:
Pre-licensure studies of GSK Biologicals' PEDIARIX vaccine have shown it to be generally safe and unlikely to result in vaccine-associated serious adverse events. This post-licensure study is designed to evaluate relatively uncommon/rare outcomes in a large population cohort.

DETAILED DESCRIPTION:
* The outcomes to be assessed include the occurrence of all seizures (with or without fever), medically-attended fever, seizures associated with fever, allergic reactions, outpatient visits and hospitalizations for any cause, and all deaths.
* Data collection through utilization of automated databases at the study site with subset medical record review. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion criteria:

Primary study cohort

The primary study cohort will include all infants from SCKP who have begun their primary course of vaccine with PEDIARIX co-administered with Prevnar and for whom at least one dose of PEDIARIX was administered prior to the infant's 9-month birthday and safety follow-up information is available.

Control cohorts

Three control cohorts will be evaluated.

1. The historical cohort will include age-, gender- and area-matched infants from SCKP who received at least one dose of DTaP vaccine co-administered with Prevnar prior to the infant's 9-month birthday and for whom safety follow-up information is available. This cohort will include infants vaccinated between January, 2002 and March, 2003.
2. The self-control cohort is defined for the study subject as the 20-day post-vaccination period from Day 21 to Day 41 for each infant in the primary cohort (PEDIARIX co-administered with Prevnar as the primary vaccination course).
3. The "delayed PEDIARIX use clinic" cohort will include all infants from SCKP who, during the enrollment period for the primary cohort, began their primary course of vaccination with DTaP vaccine and for whom at least one dose of DTaP vaccine was co-administered with Prevnar prior to the infant's 9-month birthday and safety follow-up information is available. The size of this cohort will depend on how quickly individual SCKP clinics and medical centers use PEDIARIX once it is made available. The size of this cohort, therefore, is not immediately predictable.

Exclusion Criteria: none

Ages: 6 Weeks to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will be conducted by the University of California, Los Angeles (UCLA) Center for Vaccine Research (CVR) and the Southern California Kaiser Permanente Health Care Plan (SCKP), the largest Health Maintenance Organization (HMO) in California.
  All infants who receive at least one dose of PEDIARIX in the primary series will be identified through the automated Kaiser Immunization Tracking System (KITS).
Sampling Method: Probability Sample
Enrollment: 120794 (Actual)
Dates: Start 2003-04; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
All seizures following the primary doses of PEDIARIX in Cohort A and DTaP vaccine in Cohort B | During the 8-day period following the primary dose
Medically-attended fever following the first dose of PEDIARIX in Cohort A and DTaP vaccine in Cohort B | Within 4 days following the first dose

SECONDARY OUTCOMES:
All seizures following the primary doses of PEDIARIX or DTaP vaccine | Day 21-41, in Cohort A; Day 0-7, in Cohort C
Medically-attended fever | Day 0-3 after 2nd and 3rd doses of PEDIARIX in Cohort A;Day 0-3 after 2nd and 3rd doses of DTaP vaccine in Cohort B;Day 21-41 after primary doses of PEDIARIX in the Cohort A;Day 0-3 after primary doses of DTaP vaccine in the Cohort C
Seizures associated with fever following the primary doses of PEDIARIX or DTaP vaccine | Day 0-3 after 2nd and 3rd doses of PEDIARIX in Cohort A;Day 0-3 after 2nd and 3rd doses of DTaP vaccine in Cohort B;Day 21-41 after primary doses of PEDIARIX in the Cohort A;Day 0-3 after primary doses of DTaP vaccine in the Cohort C
Allergic reactions, in cohorts A, B & C | 0 to 48 hours following the primary doses of PEDIARIX or DTaP vaccine
Outpatient visits for any cause following the primary doses of PEDIARIX or DTaP vaccine | Day 0-20, Cohort A; Day 0-20, Cohort B; Day 21-41, Cohort A; Day 0-20, Cohort C
Hospitalizations for any cause following the primary doses of PEDIARIX or DTaP vaccine | Day 0-20, Cohort A, Day 0-20, Cohort B; Day 21-41, Cohort A; Day 0-20, Cohort C
Hospitalizations for any cause following PEDIARIX or DTaP vaccine | Day 0 post dose 1 to Day 41 following the last dose and from Day 42 post last dose to 1 year following the last dose
Deaths | Day 0 post dose 1 to Day 41 following the last dose and from Day 42 post last dose to 1 year following the last dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] Zangwill KM, Eriksen E, Lee M, Lee J, Marcy SM, Friedland LR, Weston W, Howe B, Ward JI. A population-based, postlicensure evaluation of the safety of a combination diphtheria, tetanus, acellular pertussis, hepatitis B, and inactivated poliovirus vaccine in a large managed care organization. Pediatrics. 2008 Dec;122(6):e1179-85. doi: 10.1542/peds.2008-1977. PMID 19047220